CLINICAL TRIAL: NCT03601546
Title: Feasibility of Implementing a Cohort of People Living With Hepatitis C in the Viet Tiep Hospital in Hai Phong, Vietnam
Brief Title: Feasibility of Implementing a Cohort of People Living With Hepatitis C in Vietnam
Acronym: CoViet-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016-08/DL-01
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HCV infection
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination — Blood test and patient interview as for standard patient care

SUMMARY:
The purpose of this study is to evaluate the feasibility of implementing a cohort of patients with Hepatitis C in order to generate a larger cohort for future studies

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient is at least 18 years old
* The patient is HCV RNA positive

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Hepititis C recruited during consultation in the infections and tropical disease service of the Viet Tiep hospital in Hai Phong, Vietnam
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient inclusion rate | End of study: 12 months
  Number of patients included/number of eligible patients
Rate of missing data of patient variables | Day 0-1
  Current treatment, introduction of treatment, viral load, HCV genotype, fibrosis stage, HIV co-infection, drug consumption, alcohol consumption, methadone treatment,
Lost to follow-up rate | Month 6
Lost to follow-up rate | Month 12
Archival of all signed consent forms | End of study: Month 12

SECONDARY OUTCOMES:
Social-demographic characteristics of patients at inclusion | Day 0
  age, sex, weight, height, pregnancy test,
drug and alcohol consumption, | Day 0
  type and amount
treatment at inclusion | Day 0
commencement of treat | Day 1
initial HCV viral load, | Day 0
  UI/ml
HCV genotype | Day 0
Fibrosis stage | Day 0
HIV viral load | Day 0
  Copies/ml
Lymphocyte T4 level | Day 0
  Number of CD4 lymphocytes/mm3
Fibrosis stage | Day 0
  Fibroscan result
Hepatic ultrasound | Day 0
Transaminase levels | Day 0
  Gamma-glutamyl transferase, Aspartate amino transferase, Alanine amino transferase
HIV co-infection | Day 0
  Yes/no
Hepititis B co-infection | Day 0
  Yes/no
Methadone treatment | Day 0
  Yes/no
Access to health cover | Day 0
  Yes/no
Commencement of treatment | Day 1
  Yes/no
Type of treatment | Day 0
Treatment side effects | ay
Early viral response | Week 4
  Undetectable HCV RNA
Sustained viral response | Week 12
  Undetectable HCV RNA
HCV re-infection | Month 12
  Yes/no
Risk factors associated with reinfection | 3 months after clearance

CONTACTS AND LOCATIONS:
Overall Officials: Didier Laureillard, MD, Principal Investigator — CHU Nimes
Locations (2):
- CHU Nimes, Nîmes, France
- Hospital Viet Tiep, Haiphong, Vietnam